CLINICAL TRIAL: NCT06568562
Title: PRO-XL: A Phase II Study of XL092 in Patients With Metastatic Castration-Resistant Prostate Cancer After Progression on Lutetium-177 (177Lu)-PSMA-617
Brief Title: XL092 in Patients With Metastatic Castration-Resistant Prostate Cancer
Acronym: PRO-XL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI178937
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment: All Patients (Experimental): XL092 is an oral tablet that will be taken once per day on a 28 day cycle. Participants will take a 60mg dose. Dose reductions to 40mg or 20mg may apply for in cases of dose interruption due to treatment-related toxicity.
  Interventions: Drug: XL092

INTERVENTIONS:
Drug: XL092 — XL092 will be supplied as a tablet that will be taken at home once a day. Participants should drink at least 8 ounces of water with each dose of XL092. Participants should not eat at least 2 hours before taking the dose and 1 hour after. Participants will be given enough XL092 to take at home for a full cycle.
  Other Names: Zanzalintinib

SUMMARY:
The purpose of this study is to determine how well the study drug XL092 is helping to treat a participant's cancer after 16 weeks of treatment. Researchers will also look at how safe the XL092 is and how well the XL092 is working. XL092 is an oral tablet that will be taken once a day. Participants will return to clinic for regular visits for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged ≥ 18 years
* Disease criteria:

  * Histologically or cytologically confirmed prostatic adenocarcinoma without small cell histology
  * Radiographic evidence of metatstatic disease
  * Progression on or after prior treatment with 177Lu-PSMA-617 as determined by clinical investigator
* ECOG Performance Status ≤ 2.
* Adequate organ function as defined as:

  --Absolute neutrophil count ≥ 1500/mm3 .
  * Platelet count ≥ 100,000/mm3 .
  * Hemoglobin ≥ 9 g/dL .
  * Total Bilirubin ≤ 1.5x institutional ULN. For subject's with Gilbert's disease, ≤ 3 x ULN.
  * Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 3 x ULN. For subjects with documented bone metastasis ALP ≤ 5 x ULN. For subjects with CRPC and bone metastasis ALP ≤ 10 x ULN if predominantly bone-specific ALP.
  * International Normalized Ratio (INR) ≤ 1.5 and activated partial thromboplastin time (aPTT) ≤ 1.2 upper limit of normal (ULN)
  * Serum creatinine ≤ 1.5 x ULN or estimated creatinine clearance ≥ 40 mL/min by Cockcroft-Gault formula:

    ---Males: ((140-age)×weight[kg])/(serum creatinine [mg/dL]×72)
  * Urine protein-to-creatinine ratio (UPCR) ≤ 1.5 mg/mg (≤ 169.8 mg/mmol) creatinine or 24-hour urine protein <1.5 g.
* Sexually active fertile subjects and their partners must agree to use highly effective method of contraception (defined in Section 5.4.1) during the course of the study and for 96 days after the last dose of treatment (whichever is later). An additional contraceptive method, such as a barrier method (eg, condom), is required. In addition, men must agree not to donate sperm for the purpose of reproduction during these same periods.
* Must have recovered from adverse effects of any prior oncologic treatment (e.g. prior surgery, radiotherapy, or other antineoplastic therapy). CTCAE adverse events less than or equal to grade 1 are acceptable. CTCAE adverse events grade 2 or greater may be acceptable as determined by the Clinical Investigator.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Prior treatment with XL092
* Receipt of any type of small molecule kinase inhibitor, cytotoxic, biologic or other systemic anticancer therapy (including investigational) within 2 weeks or at least 5 half-lives, whichever shorter before first dose of study treatment.

Note: Concomitant use of megestrol acetate, androgen-deprivation therapy and bone loss prevention treatment is permitted. Other types of hormonal therapies with similar use require prior approval from the Principal Investigator.

* Radiation therapy for bone metastasis or any other radiation therapy within 2 weeks before first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study treatment.

Note: Subjects with an incidental finding of an isolated brain lesion < 1 cm in diameter may be eligible after Principal Investigator approval if the lesion is radiographically stable for 4 weeks before first dose and does not require treatment per Investigator judgement.

Note: Eligible subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of first dose of study treatment.

-Concomitant anticoagulation with oral anticoagulants except for those specified below:-

* (a) Prophylactic use of low-dose aspirin for cardioprotection (per local applicable guidelines), low-dose low molecular weight heparins (LMWH) or prophylactic dose of specified direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban
* (b) Therapeutic doses of LMWH or specified direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before enrollment and without clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.

  -Any complementary medications (eg, herbal supplements or traditional Chinese medicines) to treat the disease under study within 2 weeks or at least 5 half-lives, whichever shorter before first dose of study treatment.

  -The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:
* Cardiovascular disorders:

  * Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias [eg, ventricular flutter, ventricular fibrillation, Torsades de pointes (TdP)].
  * Uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic or > 90 mm Hg diastolic despite optimal antihypertensive treatment.
  * Stroke (including transient ischemic attack [TIA]), myocardial infarction, or other clinically significant ischemic event within 6 months before first dose of study treatment.
  * Pulmonary embolism (PE) or deep vein thrombosis (DVT) or prior clinically significant venous or non-CVA/TIA arterial thromboembolic events within 3 months before to first dose of study treatment.

Note: Subjects with a diagnosis of DVT within 3 months are allowed if asymptomatic and stable at screening and treated with anticoagulation per standard of care before first dose of study treatment.

Note: Subjects who don't require prior anticoagulation therapy may be eligible but must be discussed and approved by the Principal Investigator.

* Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

  ---Tumors invading the GI-tract from external viscera

  ---Active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, or acute pancreatitis

  ---Acute obstruction of the bowel, gastric outlet, or pancreatic or biliary duct within 6 months unless cause of obstruction is definitively managed and subject is asymptomatic

  ---Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose. Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose of study treatment.

  ---Known gastric or esophageal varices

  -Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 12 weeks before first dose of study treatment.
  * Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.
  * Lesions invading major blood vessel including, but not limited to, inferior vena cava, pulmonary artery, or aorta.

Note: Subjects with intravascular tumor extension (eg, tumor thrombus in renal vein or inferior V. cava) may be eligible following Principal Investigator approval.

* Other clinically significant disorders that would preclude safe study participation.

  * Active infection requiring systemic treatment. Note: Prophylactic antibiotic treatment is allowed.
  * Known infection with acute or chronic hepatitis B or C, known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
  * Known positive test for or suspected infection with clinically significant SARS-CoV-2 within one month before enrollment. Note: demonstration that the subject has fully recovered from the infection as determined by clinical investigator is required to be eligible for enrollment
  * Serious non-healing wound/ulcer/bone fracture. Note: non-healing wounds or ulcers are permitted if due to tumor-associated skin lesions.
  * Malabsorption syndrome.
  * Pharmacologically uncompensated, symptomatic hypothyroidism.
  * Moderate to severe hepatic impairment (Child-Pugh B or C).
  * Requirement for hemodialysis or peritoneal dialysis.
  * History of solid organ or allogeneic stem cell transplant.
* Major surgery (as defined in Appendix B; eg, GI surgery, removal or biopsy of brain metastasis) within 8 weeks prior to first dose of study treatment. Prior laparoscopic nephrectomy within 4 weeks prior to first dose of study treatment. Minor surgery (eg, simple excision, tooth extraction) within 10 days before first dose of study treatment. Complete wound healing from major or minor surgery must have occurred at least prior to first dose of study treatment.

Note: Fresh tumor biopsies should be performed at least 7 days before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior surgical procedures, including biopsies, are not eligible.

-Corrected QT interval calculated by the Fridericia formula (QTcF) > 480 ms for males within 14 days per electrocardiogram (ECG) before first dose of study treatment.

Note: Triplicate ECG evaluations will be performed and the average of these 3 consecutive results for QTcF will be used to determine eligibility.

* History of psychiatric illness likely to interfere with ability to comply with protocol requirements or give informed consent.
* Inability to swallow tablets.
* Previously identified allergy or hypersensitivity to components of the study treatment formulations.
* Any other active malignancy or diagnosis of another malignancy within 2 years before first dose of study treatment requiring systemic treatment, except for superficial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy.

Note: Patients with prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial as approved by the Principal Investigator.

* Other conditions, which in the opinion of the Investigator, would compromise the safety of the patient or the patient's ability to complete the study.
* Participants taking prohibited medications as described in Section 6.8. A washout period of prohibited medications for a period of at least five half-lives or as clinically indicated should occur before the start of treatment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with non-progressive disease after 16 weeks of treatment with XL092 as assessed by Prostate Cancer Working Group 3 (PCWG3)-modified RECIST v1.1 | 16 weeks
  To evaluate the disease control rate at 16 weeks in metastatic castrate-resistant prostate cancer (mCRPC) patients treated with XL092 after progression on 177Lu-PSMA-617

SECONDARY OUTCOMES:
Frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by type. | 5 years
  To evaluate the safety and tolerability of XL092 in the study population.
Frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by severity (as defined by the NIH CTCAE, version 5.0). | 5 years
  To evaluate the safety and tolerability of XL092 in the study population.
Frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by seriousness. | 5 years
  To evaluate the safety and tolerability of XL092 in the study population.
Frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by duration. | 5 years
  To evaluate the safety and tolerability of XL092 in the study population.
Frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by relationship to study treatment. | 5 years
  To evaluate the safety and tolerability of XL092 in the study population.
The proportion of patients achieving PSA decline of ≥ 50% compared to the baseline value prior to starting study treatment. | 5 years
  To evaluate the PSA 50% response rate in the study population.
Overall survival (OS) as defined as the time from study drug initiation until death from any cause. | 5 years.
  To evaluate OS in this study population.

CONTACTS AND LOCATIONS:
Overall Officials: Umang Swami, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No